CLINICAL TRIAL: NCT03374059
Title: Exercise and Life Modification Approaches for Text-Neck
Brief Title: Exercise and Life Modification for Text-Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nihan Ozunlu Pekyavas, Associated Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA 16/376
Record Dates: First submitted 2017-11-30; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Pain; Exercise; Posture
MeSH Terms: conditions — Pain; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): Exercise group received a home exercise program treatment for 4 weeks including isometric exercises for neck muscles and postural correction exercises for neck region.
  Interventions: Other: Exercise program
- Exercise and Life modification (Experimental): This group received life modification suggestions additional to home exercise treatment program for 4 weeks.
  Interventions: Other: Exercise program; Other: Life modification
- Control Group (No Intervention): Control group did not receive any treatments

INTERVENTIONS:
Other: Exercise program
  Arms: Exercise; Exercise and Life modification
Other: Life modification
  Arms: Exercise and Life modification

SUMMARY:
Objectives: The purpose of the study was to investigate the effects of exercise and life modification on pain and disability in "text neck".

Methods: Eighty-five participants were randomly divided into three groups: Exercise (n=29), Exercise+Life modification (n=28), and Control Group (n = 28). Pain intensity during rest, activity, and at night was evaluated with Visual Analogue Scale (VAS) and functional assessment was done by using Neck Disability Index at the beginning and at the end of 4 weeks.

DETAILED DESCRIPTION:
Objectives: Smartphones or tablets have made an important place in our lives. However long-term use of technological tools causes postural disorders and neck pain called "text neck". The purpose of the study was to investigate the effects of exercise and life modification on pain and disability in "text neck".

Methods: Eighty-five participants with "text-neck" were randomly divided into three groups: Exercise (n=29), Exercise+Life modification (n=28), and Control Group (n = 28). First group received a home exercise program treatment for 4 weeks. Second group received life modification suggestions additional to home exercise treatment program. Control group did not receive any treatments. Pain intensity during rest, activity, and at night was evaluated with Visual Analogue Scale (VAS) and functional assessment was done by using Neck Disability Index at the beginning and at the end of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were aged between 18 and 30, using technological devices as tablets and smartphones for more than 5 hours and having neck pain for more than 3 months were included in our study.

Exclusion Criteria:

* The exclusion criteria included those:

  1. who had any diagnosed pathology for neck region diagnosed by MR or BT,
  2. who had any shoulder pathology,
  3. with any neck or shoulder surgery,
  4. had whiplash syndrome,
  5. had fibromyalgia, Myofasial Pain Syndrome or vascular pathology and
  6. women who are breastfeeding.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 4 weeks
  Pain intensity

SECONDARY OUTCOMES:
Neck disability index | 4 weeks
  Function

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided